CLINICAL TRIAL: NCT05007860
Title: Vaccine Responsiveness in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jacob Soumerai, MD, Assistant Professor of Medicine, Clinical Investigator in Lymphoma, Massachusetts General Hospital
Other Study IDs: 20-296
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 13-valent pneumococcal vaccine; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; Ad26COVS1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No active therapy: Age ≥18 years and CLL/SLL (WHO criteria). We excluded patients with known HIV or primary immune deficiency disorder, known active progression of CLL/SLL, active therapy, treating physician intent to initiate CLL/SLL therapy within ≤2 months, prior cytotoxic chemotherapy within ≤1 year, CD20 monoclonal Ab within ≤6 months, or any prior bendamustine or fludarabine. We excluded patients who received PCV13 within ≤2 years, or within 2-5 years with nonprotective titers for ≥50% of PCV13-specific S. pneumonia IgG titers.
  Interventions: Biological: PCV13 vaccine and any of the FDA-approved COVID-19 vaccine products (BNT162b2, mRNA-1273, or Ad26.COV2.S) based on local availability.
- BTK inhibitor therapy (continued): Age ≥18 years, CLL/SLL (WHO criteria), and active therapy with a BTK inhibitor which is continued through vaccination. We excluded patients with known HIV or primary immune deficiency disorder, known active progression of CLL/SLL, prior cytotoxic chemotherapy within ≤1 year, CD20 monoclonal Ab within ≤6 months, or any prior bendamustine or fludarabine. We excluded patients who received PCV13 within ≤2 years, or within 2-5 years with nonprotective titers for ≥50% of PCV13-specific S. pneumonia IgG titers.
  Interventions: Biological: PCV13 vaccine and any of the FDA-approved COVID-19 vaccine products (BNT162b2, mRNA-1273, or Ad26.COV2.S) based on local availability.
- BTK inhibitor therapy (interrupted): Age ≥18 years, CLL/SLL (WHO criteria), and active therapy with a BTK inhibitor which is interrupted at time of vaccination. We excluded patients with known HIV or primary immune deficiency disorder, known active progression of CLL/SLL, prior cytotoxic chemotherapy within ≤1 year, CD20 monoclonal Ab within ≤6 months, or any prior bendamustine or fludarabine. We excluded patients who received PCV13 within ≤2 years, or within 2-5 years with nonprotective titers for ≥50% of PCV13-specific S. pneumonia IgG titers.
  Interventions: Biological: PCV13 vaccine and any of the FDA-approved COVID-19 vaccine products (BNT162b2, mRNA-1273, or Ad26.COV2.S) based on local availability.

INTERVENTIONS:
Biological: PCV13 vaccine and any of the FDA-approved COVID-19 vaccine products (BNT162b2, mRNA-1273, or Ad26.COV2.S) based on local availability. — Vaccines administered per standard of care

SUMMARY:
Assessment of SARS-CoV2 (mRNA and adenovirus-based vaccines) and Conjugated Pneumococcal (PCV13) in Patients with Chronic Lymphocytic Leukemia

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Age >18 years.
* Diagnosis of CLL or SLL according to WHO criteria.
* For patients receiving BTK inhibitor (Cohorts 1 and 2):

  * Patient must have no history of cytotoxic chemotherapy within 1 year (no prior history of bendamustine or fludarabine is permitted) and no history of CD20 monoclonal antibody within 6 months.
  * Patient must have no known clinical or radiographic evidence of CLL progression.
* For patients not on active therapy (Cohort 3):

  * Patient must have no history of cytotoxic chemotherapy within 1 year (no prior history of bendamustine or fludarabine is permitted) and no history of CD20 monoclonal antibody within 6 months.
  * The treating investigator must have no intention to initiate CLL therapy within 2 months.
* Patients must have not received PCV13 within 2 years. For patients with PCV13 within 5 years, S. pneumonia IgG antibody concentrations must be less than the reference value for at least 50% of S. pneumoniae serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A,19F and 23F. Patients can have received prior PPV23 within any time frame.
* Patient must have no known history of HIV or primary immune deficiency disorder, nor be taking a concurrent immune suppressing medication (e.g. steroids, methotrexate, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with CLL/SLL receiving PCV13 +/- COVID19 vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Effective immune response (EIR) to PCV13 vaccination | 35 days (+/- 14 days) after vaccination
  EIR is defined as a >2-fold increase or conversion from a nonprotective to a protective titer for >50% of specific S. pneumonia IgG titers (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) vs baseline.
Effective immune response (EIR) to COVID19 vaccination | 35 days (+/- 14 days) after vaccination
  EIR is defined as a >4-fold increase from baseline, or seroconversion defined as change from negative to within the measuring interval, for specific SARS-CoV-2 antibody titers (spike protein). For patients without pre-COVID-19 vaccination.
  serology, a negative post-COVID-19 vaccination nucleocapsid antibody titer will be used as a surrogate for no prior infection and in this case a post-COVID-19 vaccination spike antibody titer within the measuring interval will be interpreted as an EIR.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected for the study, including individual deidentified participant data and a data dictionary defining each field in the set, will be made available at study closeout.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Data will become available at study closeout and for 5 years.
Access Criteria: Request to Principal Investigator

REFERENCES:
- [Derived] Haydu JE, Maron JS, Redd RA, Gallagher KME, Fischinger S, Barnes JA, Hochberg EP, Johnson PC, Takvorian RW, Katsis K, Portman D, Ruiters J, Sechio S, Devlin M, Regan C, Blumenthal KG, Banerji A, Judd AD, Scorsune KJ, McGree BM, Sherburne MM, Lynch JM, Weitzman JI, Lei M, Kotton CN, Dighe AS, Maus MV, Alter G, Abramson JS, Soumerai JD. Humoral and cellular immunogenicity of SARS-CoV-2 vaccines in chronic lymphocytic leukemia: a prospective cohort study. Blood Adv. 2022 Mar 22;6(6):1671-1683. doi: 10.1182/bloodadvances.2021006627. PMID 35073571